CLINICAL TRIAL: NCT07258745
Title: A Randomized, Double-Blind, Single-Dose, Parallel-Group, Three-Arm Trial to Compare the Pharmacokinetics, Safety, Tolerability, and Immunogenicity Profiles of CKD-704 (Risankizumab Biosimilar), EU-approved Skyrizi®, and US-licensed Skyrizi® in Healthy Adult Participants
Brief Title: Pharmacokinetic, Safety, Tolerability, and Immunogenicity Comparison of CKD-704 (Risankizumab Biosimilar), With EU-approved Skyrizi®, and US-licensed Skyrizi® in Healthy Adult Participants
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A148_01PK2408; 2025-522345-21-00 (EU CTIS Number)
Record Dates: First submitted 2025-11-17; First posted 2025-12-02 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Psoriasis
Keywords: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — risankizumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- CKD-704 (Experimental): Singe dose pre-filled syringe, 150mg/ml
  Interventions: Biological: CKD-704
- EU-Skyrizi (Active Comparator): Singe dose pre-filled syringe, 150mg/ml
  Interventions: Biological: SKYRIZI
- US-Skyrizi (Active Comparator): Singe dose pre-filled syringe, 150mg/ml
  Interventions: Biological: SKYRIZI

INTERVENTIONS:
Biological: SKYRIZI — EU-sourced
  Arms: EU-Skyrizi
Biological: SKYRIZI — US-licensed
  Arms: US-Skyrizi
Biological: CKD-704 — Risankizumab biosimilar
  Arms: CKD-704

SUMMARY:
This is a Phase 1, first-in-human (FIH), randomized, double-blind, single-dose, parallel-group, 3-arm study to compare PK, safety, tolerability, and immunogenicity profiles of CKD-704, EU-approved Skyrizi, and US-licensed Skyrizi in healthy adult participants.

ELIGIBILITY:
Inclusion Criteria:

* Capability of giving signed informed consent and complying with the requirements and restrictions listed in the ICF and Protocol
* Healthy male or female, 18 to 55 years (inclusive) at the time of signing the ICF
* smokes ≤ 10 cigarettes per week within 3 months of screening
* abstain from alcohol from 48 hours prior to study intervention administration and keeping alcohol consumption within WHO limits (more than 14 units per week spread over 3 or more days, equivalent to 6 pints of average strength beer or 6 medium glasses [175 mL] of wine)
* have acceptable venous access for blood collection
* Female participants are eligible to participate if they are not pregnant, not breastfeeding
* Male participants must refrain from donating sperm from screening (signing the ICF) until at least 30 days after EOS visit
* All participants must be willing to use effective/highly effective methods of contraception during the study period
* Participants are willing and able to be confined to the clinical unit prior to and during the study intervention administration and required follow-up periods.

Exclusion Criteria:

* History of previous exposure to any anti-IL-12/23 or anti-IL-23 treatment
* History of relevant drug and/or food allergies
* History of hypersensitivity to Skyrizi or their constituents
* Presence of psychiatric disorders or altered mental status precluding understanding of the informed consent process and/or completion of the necessary procedures
* Medical history, findings of physical examination/laboratory tests indicate a clinically significant disorder, condition, or disease that, in the opinion of the Investigator would pose a risk to participant safety
* Major surgery within 12 weeks prior to the randomization into the study
* Documented active or suspected malignancy or history of malignancy within 5 years prior to screening
* Positive tests for hepatitis B surface antigen, Hepatitis B core antibody, hepatitis C virus antibody, or human immunodeficiency virus (HIV)-1 and HIV-2 antibody at screening
* Positive test for severe acute respiratory syndrome coronavirus 2 on admission (optional)
* Any current active infections or any recent history (within 1 week prior to study intervention administration) of active infections
* Participant has a history of tuberculosis (TB) diagnosis or evidence of active or latent infection with Mycobacterium tuberculosis
* Abnormal hepatic, renal, or hematological laboratory tests. In such cases, the assessment may be repeated once at screening and admission. The Investigator will check reassessment results to decide if the value is clinically significant and if participant is eligible to receive the treatment
* Any other laboratory value outside the reference range that the Investigator considers to be of clinical significance
* Abnormal vital signs(Systolic blood pressure < 90 mmHg or > 140 mmHg, Diastolic blood pressure < 50 mmHg or > 90 mmHg, Heart rate < 45 or > 100 beats per minute)
* Any clinically important abnormalities in rhythm, conduction, or morphology of the resting ECG and any clinically important abnormalities in the 12-lead ECG
* Any past or concurrent medical conditions, or clinically important active infection that could potentially increase the participant's risks or that would interfere with the study evaluation, procedures, or study completion
* Have used any prescription or non-prescription medicines or vitamins within 7 days or 5 half-lives (whichever is longer) of admission, unless in the Investigator's opinion will not affect determination of safety or other study assessments
* Male or females participating in any other clinical trial at the time of consenting
* Have received any investigational drug within 30 days prior to screening, with minimal washout of at least 5-half-lives of any previous investigational drug, whichever is longer
* Have received live vaccines during the past 4 weeks before screening or have the intention to receive vaccination during the 21-week treatment and assessment period
* Participant has donated blood (> 500 mL) or blood products within 2 months (56 days) prior to screening
* History of drug abuse or alcohol abuse as judged by the Investigator or designee
* Participant is affiliated with the site or Sponsor and/or may be considered to be consenting under duress
* Participant is unlikely to co-operate with the requirements of the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 213 (Estimated)
Dates: Start 2025-11-26 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Maximum Observed Serum Concentration (Cmax) | up to approximately 146 days
  Maximum observed serum concentration (Cmax) of risankizumab.
AUC From Time 0 to Infinity (AUCinf) | Up to approximately 146 days
  AUCinf of risankizumab

SECONDARY OUTCOMES:
Area Under Concentration-Time Curve (AUC) From Time 0 to Time of the Last Measurable Concentration (AUCt) | Up to approximately 146 days
  AUCt of risankizumab
Terminal Phase Elimination Hhalf-life (t1/2) | Up to approximately 146 days
  Terminal phase elimination half-life (t1/2) of risankizumab.
Time to Cmax (Tmax) | Up to approximately 146 days
  Time to Cmax of risankizumab
Safety and tolerability | Up to approximately 146 days
  Incidence and characteristics (severity, etc) of AEs

CONTACTS AND LOCATIONS:
Locations (1):
- MTZ powered by Pratia, Warsaw, Warszawa, Poland